CLINICAL TRIAL: NCT02928211
Title: An Evaluation of Aftobetin-HCl and Fluorescence Detection as Measured by Sapphire II to Determine the Number and Timing of Administrations in Subjects With Normal Cognition, Mild Cognitive Impairment, and Mild Alzheimer's Disease
Brief Title: Aftobetin-HCl and Fluorescence Detection Measured by Sapphire II to Determine the Number and Timing of Administrations
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cognoptix, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PRT-0036
Record Dates: First submitted 2016-09-19; First posted 2016-10-10 (Estimated); Last update posted 2018-08-22 (Actual); Status verified 2018-08

CONDITIONS: Mild Cognitive Impairment; Alzheimer's Disease
MeSH Terms: conditions — Cognitive Dysfunction; Alzheimer Disease | interventions — Ointments; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Experimental (Experimental): All subjects will receive the ointment and have scans with the Sapphire II device
  Interventions: Device: Sapphire II; Drug: Aftobetin-HCl; Radiation: Positron Emission Tomography

INTERVENTIONS:
Device: Sapphire II — A Class 1 laser device used in conjunction with the ointment to measure fluorescence emissions from the anterior segment (lens) of the eye.
Drug: Aftobetin-HCl — The medical imaging agent (the ointment), Aftobetin-HCl is an amyloid binding ligand formulated into an ophthalmic ointment.
  Other Names: medical imaging agent; ointment
Radiation: Positron Emission Tomography — Amyvid 370 MBq (10 mCi) is administered as a single bolus through a short intravenous catheter in a total volume of 10 mL.
  Other Names: PET

SUMMARY:
This is an open-label study to evaluate Aftobetin-HCl and florescence detection as measured by the Sapphire II device.

Performance of Part I of the study has been completed (15 subjects received a single administration of Aftobetin HCL followed by Sapphire II measurements) and indicated that 3 administrations of Aftobetin-HCl are necessary. For Part II, a second group of up to 30 subjects (CN =10 and mild AD or MCI =20) will receive three Aftobetin HCL administrations. If three administrations of Aftobetin HCL are optimal, up to an additional 30 MCI and 30 mild AD subjects will be entered.

The purpose of the study as Part II is performed is to determine the ability of the Sapphire II device to detect B-amyloid in the lens of the eye in subjects with Mild Cognitive Impairment (MCI), and mild Alzheimer's Disease (AD) after three Aftobetin-HCl administrations. Subjects with Normal Cognition (CN) will also be tested to further establish that subjects who are highly unlikely to have B-amyloid deposits in the lens of the eye will have close to baseline post ligand fluorescent uptake value (FUV) using the Sapphire II technology.

DETAILED DESCRIPTION:
Open label study. 45-105 subjects will be enrolled.

Subjects will undergo the following procedures:

* Complete physical and neurologic examination (Screening)
* Neuropsychological testing (Screening)
* Ophthalmologic examination (Screening and Visit 4 (Safety follow up visit))
* Administration of ointment - 3 administrations (Visit 1)
* Sapphire II Fluorescent Eye Measurements (Visits 1-3): Prior to first administration of ointment and then 24 +/- 2 hours, 28 +/- 30 minutes and 48 +/- 2 hours following first ointment administration
* Amyvid Positron Emission Tomography (PET) Amyloid Scan (only required for MCI and mild AD subjects who have not had a positive amyloid PET scan in the last 3 years)

Subjects will also be asked to participate in an elective second Sapphire II assessment to assess its reproducibility. Repeatability testing is optional and will require a separate consent. Subjects will come back for Visits 5-9 (ointment administration and eye scans and a follow up safety assessment).

ELIGIBILITY:
For MCI and mild AD subjects:

1. Aged 55-90 years old inclusive;
2. Able to provide informed consent;
3. Subject must have a reported memory concern verified by study partner (a study partner is someone willing to participate as a source of information and has at least weekly contact with the subject);
4. Capable of cooperating for the duration of the study with procedures and assessments;
5. Magnetic Resonance Imaging (MRI) Scan within 9 months with:

   1. Modified Hachinski Score <4
   2. No evidence of infection, infarction (ischemic or hemorrhagic), or other focal lesions (tumors, subdural hematomas, malformations, etc.)
6. Geriatric Depression Scale (GDS) score of <6;
7. Neuropsychiatric Inventory (NPI) total score <10 and <4 in any NPI domain;
8. Sufficient vision in at least one eye and hearing to participate in cognitive testing

   For MCI subjects:
9. Meets National Institute on Aging-Alzheimer's Association (NIA-AA) core clinical criteria for Mild Cognitive Impairment due to AD1;
10. Clinical dementia Rating Scale Score (CDR) of 0.5 (memory box score must = 0.5);
11. Mini-Mental State Exam (MMSE) score of >24;
12. Abnormal memory function on education adjusted Wechsler Memory Scale Logical Memory II subscale (Delayed Paragraph Recall, Paragraph A only) - Revised (16 years: <11; 8-15 years: <9; 0-7 years: <6);
13. Absence of dementia: no significant impairment in cognitive functioning or Activities of Daily Living (AODLs) - Functional Assessment Questionaire (FAQ) score of <6. The FAQ is answered by the study partner;

    For Mild AD subjects:
14. Meets National Institute on Aging-Alzheimer's Association (NIA-AA) core clinical criteria for probable AD dementia2;
15. CDR between 0.5 or 1;
16. MMSE score between 20 to 26 (inclusive);
17. Abnormal memory function on education adjusted Wechsler Memory Scale Logical Memory II subscale -(Delayed Paragraph Recall, Paragraph A only) -Revised (16 years: <8; 8-15 years: <4; 0-7 years: <2);
18. Functional Assessment Questionaire (FAQ) score of >6. The FAQ is answered by the study partner;

    For CN subjects:
19. Subject must be free of memory complaints;
20. Cognitively normal, based on an absence of significant impairment in cognitive functions or activities of daily living;
21. Normal memory function documented by scoring above education adjusted cut-offs on the Logical Memory II subscale (Delayed Paragraph Recall, Paragraph A only) from the Wechsler Memory Scale - Revised (≥11 for 16 or more years of education; ≥9 for 8-15 years of education;
22. MMSE score of 29-30;
23. CDR Scale Score of 0;
24. Aged 25-40 years old inclusive; and
25. Negative family history for onset of memory dysfunction in first or second degree relatives before age 65.

Exclusion Criteria:

1. Serious underlying medical disease which in the opinion of the investigator may interfere with the participant's ability to participate in the study such as unstable cardiac, pulmonary, renal, hepatic, endocrine, hematologic, active malignancy or infectious disease;
2. Non-AD causes of dementia that could cause impaired memory ruled out by standardized work up for dementia;
3. Significant neurologic disease (e.g., Parkinson's Disease, Huntington's disease, normal pressure hydrocephalus, brain tumor, progressive supranuclear palsy, seizure disorder, subdural hematoma, multiple sclerosis);
4. Clinically relevant, abnormal serum chemistry, B12, TSH, and CBC <6 months of study entry;
5. History of significant head trauma followed by persistent neurologic defaults or known structural brain abnormalities, learning disability or mental retardation;
6. Significant psychiatric illness in last year such as major depression, bipolar, obsessive compulsive or psychotic disorder;
7. History of alcohol or substance abuse in last year;
8. Pain or sleep disorder that could interfere with cognitive testing;
9. Known hypersensitivity to Amyvid (Florbetapir-F 18) or any components of injection formulation or contraindication to PET scan (e.g., pregnant, lactating, or of childbearing potential) in subjects requiring a PET scan.
10. Receiving any investigational medications or participated in a trial with investigational medications within 30 days prior study entry;
11. History of bilateral cataract surgery;
12. Active ocular inflammation or infection;
13. History of physical injury or other serious eye disease;
14. Corneal disease that prevents visualization of the lens, e.g, Fuch's dystrophy or keratokonus;
15. Inability to tolerate the PET environment, e.g., due to physical size and/or claustrophobia in subjects requiring a PET scan.
16. Serious suicidal ideation in the opinion of the investigator or answers 'yes' to Item 4 or 5 on the Columbia Suicide Severity Rating Scale (CSSRS) at screening;
17. Inability to undergo MRI procedure (e.g., metal implant, metallic devices, e.g., non-MRI-safe cardiac pacemaker or neuro-stimulator, some artificial joints, metal pins, surgical clips, other implanted metal, or claustrophobia or discomfort in confined spaces)
18. May not be taking any of the following psychoactive medications:

    * Regular use narcotic analgesics (>2 doses/ week)
    * Clonidine, neuroleptics, antidepressants with central anticholinergic activity
    * Other agents with central anticholinergic activity such as diphenhydramine, hydroxyzine, benztropine
    * Diazepam, clonazepam, temazepam, chlordiazepoxide, or triazolam

Note: it is permitted to remain on the following psychoactive medications provided the subject has been receiving them for greater than or equal to 4 weeks:

* Antidepressants lacking significant anticholinergic side effects
* Estrogen replacement therapy
* Gingko biloba
* Sedative hypnotics: lorazepam, buspirone, oxazepam, zolpidem, zaleplon, alprazolam, chloral hydrate

Note: it is permitted to remain on the following psychoactive medications provided the subject has been receiving them for greater than or equal to 12 weeks:

* Cholinesterase inhibitors
* Memantine Note: the washout from psychoactive medication (e.g., excluded antidepressants, neuroleptics, chronic anxiolytics or sedative hypnotics) must be at least 4 weeks prior to screening.

Ages: 25 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 105 (Estimated)
Dates: Start 2016-07 (Actual); Primary Completion 2018-12 (Estimated); Study Completion 2019-01 (Estimated)

PRIMARY OUTCOMES:
Paired pre-ligand and post ligand fluorescent uptake values (FUV) | through study completion, approximately 4 weeks
Determination of success (yes or no) | through study completion, approximately 4 weeks
  Determination of success (yes or no) associated with FUVs obtained after one dose or two doses of ligand at each time point by subject
The overall diagnostic precision for each combination of Aftobetin-HCl administrations and Fluorescent Uptake Value (FUV) | through study completion, approximately 4 weeks
  The overall diagnostic precision for each combination of:
  * The number of Aftobetin-HCl administrations and
  * Fluorescent Uptake Value (FUV): amyloid binding of Aftobetin-HCl to the lens of the eye as measured by Sapphire II system at 1, 2, 3, 4, 5, 6 (+/-10 minutes) and 24 hour (+/- 2 hours) time points for Part I and
  * Fluorescent Uptake Value (FUV): amyloid binding of Aftobetin-HCl to the lens of the eye as measured by Sapphire II system at 24 hours (+/-2 hours), 28 hours (+/- 30 minutes) and 48 hours (+/- 2 hours) for Part II.

SECONDARY OUTCOMES:
Estimates of sensitivity and specificity of MCI and mild AD subjects compared to cognitively normal subjects | through study completion, approximately 4 weeks
Safety of Sapphire II procedure as determined by instances of Adverse Events | through the follow up safety visit, approximately 4 weeks
Characterization of maximal fluorescence after 1, or potentially 3, ointment administrations | through study completion, approximately 4 weeks
Intra-class correlation of the repeatability of the Sapphire II measurements to verify the system's reliability for reproducible results | through study completion, approximately 6 weeks
  Optional repeatability portion of the study
Correlation of FUV to PET amyloid status | through study completion, approximately 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Joyce Myers, MD, Study Director — Cognoptix, Inc.
Locations (1):
- Neurology Research Institute, West Palm Beach, Florida, United States

IPD SHARING:
Plan to Share IPD: Yes
Subjects will receive copies of their PET scans following completion of their participation in the study